CLINICAL TRIAL: NCT06307587
Title: Vastus Intermedius Dry Needling for Knee Stiffness Resulted From Surgically Managed Femoral Fractures With Open Reduction & Internal Fixation; Randomized Controlled Trial (ORIFDN Trial)
Brief Title: Vastus Intermedius Dry Needling for Knee Stiffness Resulted From Surgically Managed Femoral Fractures With Open Reduction & Internal Fixation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Razi Hospital (Other Government)
Responsible Party: Principal Investigator, Najla Alsiri, Principal Investigator, Al-Razi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/2355
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DN group (Active Comparator)
  Interventions: Procedure: dry needling
- Control group (No Intervention)

INTERVENTIONS:
Procedure: dry needling — The vastus intermedius will be approached with DN from the lateral aspect and the pincer approach will be followed. The Hong fast-in and fast out technique with multiple rapid needle insertions will be performed following previous recommendations (Chou, et al., 2014). The control group will receive the rehabilitation program alone. A headless 0.25 × 25-mm needle (Stainless steel, Agupunt A1038P, 158 Caspe, Barcelona, Spain) will be used. The penetration depth will be varied according to the patient. Hemostasis will be performed for 1 minutes. DN will be performed medial to the sartorius muscle limit to avoid saphenous nerve adverse effects during DN (Henry et al., 2016).
  Arms: DN group

SUMMARY:
Orthopedic traumatic injuries are considered a major health epidemic, challenged by high morbidity, mortality, and socioeconomic burden. The management of traumatic orthopedic injuries is challenging and complex, with high resources utilization. Particularly, the prevalence of femoral fractures in Kuwait is 8.8%, being one of the most prevalent injuries. Open reduction and internal fixation (ORIF) is a common surgical procedure for the management of femoral fractures demonstrating successful outcome for allowing minimally invasive percutaneous plate osteosynthesis, early union of 93% to 100%, and low infection rate of only 0% to 2%. Yet, one of the major complications post ORIF is knee stiffness and reduced function, which brings many inconveniences to patients' daily lives, lead to disability, and could seriously threaten the functional activities of patients. The incidence of knee stiffness requiring surgical intervention is 14.5%. Particularly, the potential loss of knee flexion is 30 to 40 degrees, 13% of the patients failed to reach 90 degrees of knee flexion, and only 48% of patients reached >120 degrees of flexion. Ultimately, knee stiffness in flexion forms a major issue in distal femoral fractures. Various reasons could explain such complication including intrinsic adhesions, fibrosis and shortening of the vastus intermedius muscle.

There are various surgical procedures which could be used to manage knee stiffness. However, there is no consensus regarding the ideal approach and strategy with many postoperative complications including deep sepsis, quadricep tendon rupture, skin dehiscence and infection, delayed wound healing, patella fracture, lateral femoral condyle fracture and extension lag. In contrast, dry needling (DN) is a minimal invasive intervention for the management of musculoskeletal dysfunction, and it could be used to reduce the adhesion and fibrosis between the vastus intermedius and the femoral bone. However, there is limited research investigating the effect of DN on the vastus intermedius muscle after ORIF of the femoral fractures. The effectiveness of DN was explored for the management of various musculoskeletal conditions, and a systematic review addressing DN in the lower quarter concluded that DN is an effective procedure (Morihisa et a,., 2016). In ACL reconstruction, DN for the vastus medialis improved ROM at short-term and improved function at both short and long term. DN has been proposed as a useful addition to the rehabilitation of ACL reconstructed in reducing pain intensity, increasing knee flexion range, and modifying the mechanical properties of the quadriceps muscle during the late-stage of rehabilitation. DN has also altered the passive mechanical properties of the quadriceps muscle where decrement and resistance of the vastus medialis were significantly reduced. It is hypothesized that releasing the adhesions and fibrosis of the vastus intermedius could play an important role in managing knee stiffness post ORIF of the distal femur fractures. Therefore, the aim of this project is to identify the incidence rate and risk factors of knee stiffness resulted from surgically managed femoral fractures with open reduction and internal fixation in Kuwait, and to investigate the effect of DN on the vastus intermedius muscle in improving knee joint range of motion and function after ORIF of the distal femur using single blind randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55-year-old participants.
* Distal one third femur fractures classified as type 33 with AO/OTA classification.
* Three months post ORIF surgery to the distal femoral fracture,
* Experience postoperative limitation in knee flexion range of motion of less than 90 degrees.

Exclusion Criteria:

* Neuropathic pain in the lower limb.
* Lumbosacral radiculopathy,
* Saphenous nerve entrapment,
* Meralgia paresthetica,
* Rheumatoid or systemic conditions,
* Other surgeries,
* Post-surgery complications (i.e., thrombosis or osteomyelitis) or use of heparin during DN.
* Knee surgery,
* Periprosthetic fractures,
* Scraw fixation only,
* Intermedullary nail fixation,
* non-union,
* Isolated medial or lateral condyle femoral fractures,
* Underwent manipulation under anesthesia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-12 (Estimated)

PRIMARY OUTCOMES:
knee flexion range of motion | one month, 6 months, 12 months
  Knee flexion range of motion will be the primary outcome measure, which will be measured with standard goniometry in supine position considering the lateral femoral epicondyle as the center of the fulcrum. Knee extension will also be measured in supine position.

IPD SHARING:
Plan to Share IPD: No